CLINICAL TRIAL: NCT02755896
Title: Prone Partial Breast Irradiation (PBI): Prospective Randomized Controlled Non-inferiority Trial to Compare Radiation Fibrosis With Five Versus Three Fractions
Brief Title: Trial to Compare Radiation Fibrosis With Five Versus Three Fractions
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1505016201
Record Dates: First submitted 2015-08-27; First posted 2016-04-29 (Estimated); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasm of Breast Stage I
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Arm 1 - 600 cGY x 5 fractions (Other): Patients will receive 600 cGY x 5 fractions of radiation therapy over 5 consecutive days.
  Interventions: Radiation: Arm 1 600 cGY x 5 fractions
- Arm 2 - 800 cGY x 3 fractions (Other): Patients will receive 800 cGY x 3 fractions of radiation therapy every other day for 3 days.

INTERVENTIONS:
Radiation: Arm 1 600 cGY x 5 fractions — Patients who are randomized to Arm 1 will receive either 600 cGY x 5 fractions over 5 consecutive days
  Arms: Arm 1 - 600 cGY x 5 fractions
Radiation: Arm 2 800 cGY x 3 fractions — Patients who are randomized to Arm 2 will receive 800 cGY x 3 fractions given every other day

SUMMARY:
Post meno-pausal women with T1 Breast cancers will be randomized to receive either 600 centiGray (cGy) X 5 over five consecutive days (arm 1) versus 800 cGy X 3 fractions given every other day (arm 2). Patients will complete treatment in one week. All patients will be followed a month after the completion of treatment then q6 months for the first year, then yearly for the next 10 years.

DETAILED DESCRIPTION:
Partial breast irradiation (PBI) is becoming a new paradigm for breast cancer radiation. No type I or II evidence is currently available to demonstrate equivalence to standard whole breast radiotherapy, and a prospective randomized trial jointly sponsored by NSABP and Radiation therapy Oncology Group (RTOG) (NSABP B-39 and RTOG 0413) has completed accruing patients, comparing whole breast radiotherapy to PBI, either by brachytherapy or external beam techniques (EB): results of this trial are pending. Until results of this or similar trials are available, PBI remains a research domain, and it should be offered to patients only in the context of a clinical experimental protocol. Despite the fact that less extensive experience than that of brachytherapy is available, PBI delivery through an external-beam has many advantages. First of all, it is likely to be more acceptable to the patient since it is non-invasive and it does not require a surgical procedure or anesthesia. Moreover, since it is delivered after surgery, the pathological analysis of the segmental mastectomy specimen is available to inform the selection of the best candidates. In addition, EB-PBI is likely to become more widely reproducible, since it does not rely on the experience and skills of the radiation oncologist performing the brachytherapy implant. Besides, once the technique is established, it can be widely applied at any facility provided with a linear accelerator, without the risk presented by some brachytherapy approaches that cannot be completed because of the unfavorable interplay of patient's anatomy with the technical limitations of the applicator. Finally, in terms of health care economics, an external beam approach spares the costs of an extra surgical procedure and several days as inpatient (in the case of Low dose Rate (LDR) brachytherapy).

A prone approach for partial breast radiation has been tested at NYU in a clinical trial sponsored by an IDEA grant of the Department of Defense (NYU 00-23). Results of the first 47 patient accrued originally demonstrated feasibility. Eligibility to this study was limited to post-menopausal women with non-palpable, mammographically detected tumors. In addition, the protocol required patients to have first refused to undergo standard six-week radiotherapy. Five fractions of 6 Gy were delivered to the Planning Target Volume (PTV) over ten days (Monday-Wednesday-Friday, Monday-Wednesday). The dose and fractionation was based on radiobiological modeling, aimed at determining a dose to deliver in five fractions that would achieve equivalence to the tumor control estimates of 50 Gy in 25 fractions, while maintaining a risk of fibrosis at the tumor bed comparable to that of a standard regimen of 60 Gy in 30 fractions. An α/β = 4 for tumor control was used, and its validity has been recently confirmed by the results of a prospective randomized trial comparing accelerated to standard whole breast radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Post-menopausal women with status post segmental mastectomy defined as either 1) at least 2 years without menstrual period or 2) or patients older than 50 with serological evidence of post-menopausal status or 3) hysterectomized patients of any age with Follicle Stimulating Hormone (FSH) confirmation of post-menopausal status.
2. Stage 1 (pT1) breast cancer, excised with negative margins.
3. clinically N0 or No Regional Lymph node (pN0) or sentinel node negative

Exclusion Criteria:

1. Previous radiation therapy to the ipsilateral breast.
2. Presence of a proportion of Ductal Carcinoma in-situ (DCIS) in the core biopsy specimen which is compatible with extensive intraductal component (EIC).

Ages: 50 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2015-10-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with grade 2 or 3 fibrosis between the two treatment groups will be compared. | 60 months
  The primary analysis will be the difference in proportions of patients with grade 2 or 3 fibrosis between the two treatment groups compared using a non-inferiority z- test. The proportions of patients by grade of fibrosis will be compared in the two treatment arms using contingency table methods and chi square tests.

SECONDARY OUTCOMES:
Recurrence rates will be documented | 60 months
  Rates of recurrence at 1, 2, and 3 years post-randomization will be estimated with 95% confidence limits within treatment groups along with plots of Kaplan-Meier time to recurrence curves

CONTACTS AND LOCATIONS:
Overall Officials: Silvia C Formenti, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (4):
- United States (4):
  - University of Southern California, Los Angeles, California
  - Weill Cornell Medical College, New York, New York
  - Brooklyn Methodist Hospital - NewYork Presbyterian, New York, New York
  - New York Presbyterian Hospital - Queens, New York, New York

IPD SHARING:
Plan to Share IPD: No
All data and medical information obtained will be kept confidential to the extent permitted by law and will not be released without the patient's written permission except as described in this paragraph. In all study forms, patients will be identified only by their initials and patient number. Patient names will not be reported in any publication; only the data obtained as a result of their participation in this study will be made public.